CLINICAL TRIAL: NCT06935643
Title: The Effect of Birth Ball and Perineal Massage on Perineal Pain, Perineal Trauma and Birth Satisfaction During the Intrapartum Period
Brief Title: The Effect of Birth Ball and Perineal Massage on Perineal Pain, Perineal Trauma and Birth Satisfaction
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, İrem Altun, Master Student, Istanbul University - Cerrahpasa
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: IUC-EBE-IA-01
Record Dates: First submitted 2025-03-31; First posted 2025-04-20 (Actual); Last update posted 2025-04-24 (Actual); Status verified 2025-04

CONDITIONS: Perineal Pain; Birth Satisfaction; Perineal Laceration, Tear, or Rupture During Delivery
Keywords: Birth Satisfaction; Perineal trauma; Birth Ball; The Effect of perineal massage; The Effect of birth ball
MeSH Terms: conditions — Lacerations | interventions — Control Groups

STUDY DESIGN:
Intervention Model Description: In the study with 3 groups, there were perineal massage group, birth ball group and control group.
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Birth Ball Group (Active Comparator): The use of a birth ball is a non-pharmacological method to reduce labor pain is one of the methods. It is a low-cost and reliable method of dealing with pain. Birth balls of different sizes and shapes such as Swiss ball, bean-shaped, peanut-shaped are used. The birth ball , which is usually 55 cm or 65 cm in diameter, is round and plastic. Sitting on the birth ball, rocking and pelvic rotation movements reduce pain in pregnant women and facilitate labor.
  Interventions: Other: Birth Ball
- Perineal Massage Group (Active Comparator): Perineal massage; It is a safe method of preventing perineal trauma. As a result of studies on the use of liquid petroleum jelly for perineal massage application, the importance of vaseline perineal massage in preventing the development of trauma has been emphasized. Thanks to the lubricating effect of liquid petroleum jelly, it has been observed that the risk of developing perineal trauma is reduced
  Interventions: Other: Perineal Massage
- Control Group (Active Comparator): Pregnant women in the control group will be given routine midwifery care without any intervention.
  Interventions: Other: Control Group

INTERVENTIONS:
Other: Birth Ball — Written and verbal consent will be obtained by giving information about the study.The Pregnant Diagnosis Form will be filled out.When the cervical opening is 4-5 cm, 6-7 cm and 8-10 cm, the pregnant woman will have a birth ball application for 10 minutes. Visual Analog Scale (VAS) will be completed before and after each application. During labor, the Labor Monitoring and Perineal Trauma Assessment Form will be completed and the presence/degree of perineal trauma will be evaluated.Visual Analog Scale (VAS) will be completed at the 1st hour postpartum.At the 4th hour postpartum, the Visual Analog Scale (VAS) and The Scale for Measuring Maternal Satisfaction in Birth will be completed.
  Arms: Birth Ball Group
Other: Perineal Massage — Written and verbal consent will be obtained by giving information about the study.The Pregnant Diagnosis Form will be filled out. When the cervical opening is 4-5 cm, 6-7 cm and 8-10 cm, 10 minutes of perineal massage will be applied to the pregnant woman. Visual Analog Scale (VAS) will be completed before and after each application. During labor, the Labor Monitoring and Perineal Trauma Assessment Form will be completed and the presence/degree of perineal trauma will be evaluated.Visual Analog Scale (VAS) will be completed at the 1st hour postpartum.At the 4th hour postpartum, the Visual Analog Scale (VAS) and The Scale for Measuring Maternal Satisfaction in Birth will be completed.
  Arms: Perineal Massage Group
Other: Control Group — Pregnant women in the control group will not receive any intervention. Pregnant women in this group will only receive routine midwifery care.
  Written and verbal consent will be obtained by giving information about the study.Pregnancy Diagnosis Form will be filled.When the cervical opening is 4-5 cm, 6-7 cm and 8-10 cm, Visual Analog Scale (VAS) will be completed. During labor, the Labor Monitoring and Perineal Trauma Assessment Form will be completed and the presence/degree of perineal trauma will be evaluated.Visual Analog Scale (VAS) will be completed at the 1st hour postpartum.At the 4th hour postpartum, the Visual Analog Scale (VAS) and The Scale for Measuring Maternal Satisfaction in Birth will be completed.
  Arms: Control Group

SUMMARY:
One of the important causes of perineal trauma is perineal tension. By reducing this tension, perineal trauma can be prevented. Perineal trauma is a birth complication that can be prevented with midwifery approaches. The aim of this study was to investigate the effect of birth ball and perineal massage on perineal pain, perineal trauma and labor satisfaction in the intrapartum period.

DETAILED DESCRIPTION:
Perineal trauma is the disruption of perineal integrity that develops in the genital area at birth and occurs spontaneously or as a result of surgical intervention. One of the important causes of perineal trauma is perineal tension. Perineal traumas can be prevented by reducing this tension.Birth ball and perineal massage are recommended approaches to prevent perineal trauma from the active phase. As a result of these approaches, an increase in birth satisfaction, an increase in quality of life, a decrease in perineal pain and continuity of communication between mother and baby are provided.Massage is started by applying a lubricant to the hands and the fingers are placed into the vagina until the first knuckle. The thumb and index fingers are moved in a "U" shape by pressing the rectum and the tension of the perineal muscles is reduced. In the Positive Birth Experience Booklet published by the World Health Organization, it recommends perineal massage in the second stage of labor to facilitate vaginal delivery and reduce perineal trauma. At a high level of evidence, perineal massage is recommended to prevent third and fourth degree perineal trauma. Perineal trauma care is a condition that increases the cost of delivery, and perineal massage reduces the cost of care and provides quality midwifery care.The use of a birth ball in the intrapartum period increases uterine blood flow, relaxes the muscles and thus reduces pain. Its use is recommended because of its effects on the birth process such as completing the engagement of the fetal head, shortening the duration of the latent phase and increasing the comfort of labor. In addition, the movement of the mother on the birth ball increases the flexibility of the perineal muscles and reduces the risk of perineal trauma. The use of a birth ball is recommended in the first and second stages of labor.

ELIGIBILITY:
Inclusion Criteria:

* Between 18-35 years old
* Active phase
* Multipar
* Singleton pregnancy
* No risky pregnancy
* No complications for vaginal delivery
* Gestational week between 37-42
* The amniotic membrane has not opened
* No perineal scar tissue
* The anterior cephalic position of the fetal head
* Can speak and understand Turkish
* Pregnant women who agreed to participate in the study

Exclusion Criteria:

* Macrosomic fetus (birth weight over 4000 grams according to ultrasound calculation)
* Vaginal infection and/or sexually transmitted disease

Research Termination Criteria

* Cesarean section decision following trauma (due to fetal distress etc.)
* Pregnant women who develop complications during labor (instrumental delivery, etc.)
* Pregnant women who wish to withdraw from work

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 144 (Estimated)
Dates: Start 2025-05-01 (Estimated); Primary Completion 2025-10-01 (Estimated); Study Completion 2025-10-01 (Estimated)

PRIMARY OUTCOMES:
Perineal Pain Assessment | Cervical dilatation will assses is 4-5 cm, 6-7 cm ve 8-10 cm until delivery. Pain will be evaluated at the 1st and 4th hour after delivery.
  The Visual Analog Scale (VAS) is a scale used to measure pain and other subjective symptoms. It was first introduced by Hayes and Patterson in 1921. The scale has a maximum score of 10 and a minimum score of zero. And as the scale score increases, the measure of pain also increases. High scores indicate severe pain, while low scores indicate reduced pain. When cervical dilatation is 4-5 cm, 6-7 cm and 8-10 cm, the pregnant woman is asked to mark the pain score from one to ten on the VAS (Visual Analog Scale) score, and then massage is applied for 10 minutes.
Perineal Trauma Assessment | Perineal trauma will be assessed within 1 hour after birth.If the trauma has developed, it is marked as 'developed'; if the trauma has not developed, it is marked as 'not developed'.
  The Labor Monitoring and Perineal Trauma Assessment Form, prepared by the researcher in line with the literature, consists of 24 questions that question information about labor, the presence/degree of perineal trauma and information about the newborn. Perineal trauma will be evaluated by considering the recommendations of the International Incontinence Association and RCOG (2015). The form will be completed by the researcher during labor.
Assessing Maternal Satisfaction at Birth | At the 4th hour after birth, maternal satisfaction will be assess.As the total score obtained from the scale increases, the satisfaction levels of mothers regarding the care they receive in the hospital during normal childbirth also increase.
  Developed in 2009 by Güngör and Beji, the Maternal Satisfaction in Childbirth Assessment Scale is a 5-point Likert-type scale consisting of 43 items and 10 sub-dimensions. The sub-dimensions of the scale are perception of the health care team, nursing care during the birth process, comfort, participation in decisions and information, meeting her baby, care in the postpartum period, hospital room, hospital facilities, respect for privacy and meeting expectations. the Maternal Satisfaction in Childbirth Assessment Scale is applied to women who have just given birth.The sum of the scores of all items in the scale gives the "total scale score". The total raw score ranges from 43-215. As the total score obtained from the scale increases, the satisfaction levels of the mothers with the care they receive in the hospital during normal birth increase. The point score calculated for the Maternal Satisfaction Assessment Scale in Normal Birth was determined as 150.5 (≥150.5 sThe cronbach alpha va

IPD SHARING:
Plan to Share IPD: No